CLINICAL TRIAL: NCT05990608
Title: The Validity and Reliability of The Peabody Developmental Motor Score In Children With Preschool Duchenne Muscular Dystrophy
Brief Title: Peabody Developmental Motor Scaling In Children With Period Duchenne Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Deniz Çakır, Research Assistant, Ondokuz Mayıs University
Other Study IDs: 2021/371
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy (DMD); Peabody Developmental Motor Scales-2
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Healthy Children
  Interventions: Other: Peabody Developmental Motor Scales-2, PDMS
- Group II: Children with DMD
  Interventions: Other: Peabody Developmental Motor Scales-2, PDMS

INTERVENTIONS:
Other: Peabody Developmental Motor Scales-2, PDMS — The Peabody Developmental Engine Scales-2, PDMS, is a standardized norm-referenced test used to determine the motor skill level of children aged 0 to 6, identify delays in engine development, and determine individual needs and challenges. The 2 scalar, which allows children to evaluate rough and thin motor skills, consists of 6 sub-tests and 249 articles. The rough motor scale contains 4 sub-tests and 151 items, including reflex, equilibrium, locomotion and object manipulation. The slim motor scale consists of 2 sub-tests and 98 items, including cognition and visual-motor integration. Using the age-appropriate normal value ranges in the test manual to determine developmental stress risk and level, the coarse motor skills, slim motor skills, and general motor development are categorized as "very low, low, below average, above average, high, very high".

SUMMARY:
To perform the reliability and validity study of the Peabody Developmental Motor Scale (Peabody Developmental Motor Scales-2) in children with Duchenne Muscular Dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

* for Group I:

  * No neurodevelopmental problems or diseases
  * 3-5 years old
  * Being able to cooperate with the instructions given by the physiotherapist.
  * Children who volunteered to participate in the study and whose families gave consent form will be included in the study.
* for Group II:

  * Being diagnosed with Duchenne Muscular Dystrophy by a pediatric neurologist
  * 3-5 years old
  * Children who volunteered to participate in the study and whose parents' consent was obtained will be included in the study.

Exclusion Criteria:

* Children with a behavioral condition and any disorder that interferes with testing (eg autism spectrum disorder)
* Failure to cooperate with the physiotherapist who made the evaluations.
* Lack of volunteers.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Ondokuz Mayıs University, Health Application and Research Center, Pediatric Neurology Outpatient Clinic and community samples
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales-2 | This assessment will take place over the course of the study started and to the finish time

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Çakır, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No